CLINICAL TRIAL: NCT03892434
Title: Bevacizumab Versus DEX Implant Followed by Bevacizumab in ME Secondary to BRVO
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yeungnam University College of Medicine (Other)
Responsible Party: Principal Investigator, Min Sagong, Associate Professor, Yeungnam University College of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: YUMC 2019-02-018
Record Dates: First submitted 2019-03-26; First posted 2019-03-27 (Actual); Last update posted 2019-03-27 (Actual); Status verified 2019-03

CONDITIONS: Branch Retinal Vein Occlusion With Macular Edema
MeSH Terms: interventions — Dexamethasone

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Bevacizumab (Active Comparator)
  Interventions: Drug: Intravitreal bevacizumab and dexamethasone implant Injection
- Dexamethasone (Active Comparator)
  Interventions: Drug: Intravitreal bevacizumab and dexamethasone implant Injection; Device: Intravitreal dexamethasone implant

INTERVENTIONS:
Drug: Intravitreal bevacizumab and dexamethasone implant Injection — Bevacizumab 1.25mg is injected into the vitreous cavity through the pars plana using 30G needle-attached syringe for branch retinal vein occlusion, and Dexamethasone 0.75mg implant is injected using injector.
  Other Names: Intravitreal dexamethasone implant
Device: Intravitreal dexamethasone implant — Dexamethasone implant insertion using approved kit
  Arms: Dexamethasone

SUMMARY:
To evaluate the efficacy of sequential therapy with intravitreal dexamethasone implant followed by bevacizumab compared with bevacizumab monotherapy for macular edema (ME) secondary to retinal vein occlusion (RVO).

DETAILED DESCRIPTION:
Retinal vein occlusion is the second most common retinal vessel disease following diabetic retinopathy. It is divided into central retinal vein occlusion and retinal vein occlusion. Visual disturbance resulting from retinal vein occlusion is mainly caused by macular edema, and one of the main mechanisms of macular edema is increased vascular endothelial growth factor. Increased vascular endothelial growth factor is known to cause macular edema by breaking blood retinal barrier and causing leakage. For this reason, intravitreal injection of anti - vascular endothelial growth factors is currently used to treat macular edema due to retinal vein occlusion. Corticosteroid is a different mechanism from anti - vascular endothelial growth factor, and it is the main mechanism to suppress macular edema, to suppress the expression of inflammatory mediators, to block the inflammatory reaction pathway, and to lower the vascular endothelial growth factor concentration in the vitreous body. The dexamethasone implant in the vitreous cavity showed the maximum visual improvement effect during 60 day after one injection, and the effect continued until about 90 days after the injection. The same effect was obtained with a fewer injection times compared to the injection of the anti-vascular endothelial growth factor and a variety of inflammatory. It is also effective in patients who do not respond to anti-vascular endothelial growth factors by effectively inhibiting cytokines and growth factors. However, steroids elevated intraocular pressure, it is limited in repeated use.

Intravitreal dexamethasone implantation and anti-vascular endothelial growth factor showed similar early vision improvement. The differences in these anatomical changes may be different in long-term visual prognosis. After 3 doses of loading dose of anti-vascular endothelial growth factor, each group was injected with anti-vascular endothelial growth factor (VEGF) at each recurrence of macular edema and injected with anti-vascular endothelial factor at each macular reattachment after dexamethasone injection. The results of this study are as follows.

ELIGIBILITY:
Inclusion Criteria:

Center-involved macular edema secondary to BRVO for no longer than 3 months (at the screening visit it should be ensured that the subjects will comply with the criterion of ≤ 3 months since onset of macular edema at their scheduled baseline visit).

Exclusion Criteria:

* Previous PRP or macular laser photocoagulation in the study eye.
* Any prior or concomitant ocular treatment (e.g. anti-VEGF therapy, corticosteroids) in the study eye for macular edema secondary to BRVO, except dietary supplements or vitamins prior to inclusion in the study. Intraocular anti-VEGF treatment is permitted for the treatment of diseases of fellow eye except for those that are specifically excluded.
* Prior systemic anti-VEGF or corticosteroid therapy, investigational or approved, within the last 3 months before the first dose in the study.
* Previous use of intraocular corticosteroids in the study eye at any time or use of periocular corticosteroids in the study eye within 12 months prior to Day 1.
* Any active intraocular, extraocular, and periocular inflammation or infection in either eye within 4 weeks of screening.
* Any history of allergy to povidone iodine.
* Known serious allergy to the fluorescein sodium for injection in angiography.
* Presence of any contraindications indicated in the EU commission/locally approved label for intravitreal aflibercept: hypersensitivity to the active substance intravitreal aflibercept or to any of the excipients; active or suspected ocular or periocular infection; active severe intraocular inflammation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-03-18 (Actual); Primary Completion 2019-12-18 (Estimated); Study Completion 2020-06-18 (Estimated)

PRIMARY OUTCOMES:
Mean change of best corrected visual acuity | From baseline to Week 24
  The mean change of best corrected visual acuity from baseline to Week 24 in Snellen visual acuity

CONTACTS AND LOCATIONS:
Locations (1):
- Yeungnam university hospital, Daegu, South Korea

IPD SHARING:
Plan to Share IPD: No